CLINICAL TRIAL: NCT01409304
Title: Effectiveness of Deep Transcranial Magnetic Stimulation for Treating Major Depression: a Pilot Study
Brief Title: Effectiveness of Deep Transcranial Magnetic Stimulation in Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, MARCELO T. BERLIM, Director, Neuromodulation Research Clinic, Douglas Mental Health University Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTMS-ERB10/18-2011
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Major Depressive Disorder
Keywords: Major depression; Deep Transcranial Magnetic Stimulation; Naturalistic Trial; DTMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation (DTMS) — DTMS will be administered according to the following parameters: 18 Hz in 84 trains of 2 seconds duration, with 20 seconds inter-train interval (3,024 pulses per session) at 120% of the resting motor threshold.

SUMMARY:
We intend to investigate whether deep transcranial magnetic stimulation (DTMS), a novel brain stimulation technique, is effective for treating major depression. We hypothesize that 4 weeks of DTMS will be associated with significant improvements in depressive and anxious symptoms without significant side effects.

DETAILED DESCRIPTION:
The aim of this pilot study is to assess, naturalistically, the effectiveness of deep transcranial magnetic stimulation (DTMS) in a sample of subjects with treatment-resistant depression. To do this, enrolled depressed outpatients will be assigned to receive 4 weeks of daily DTMS and will be evaluated at baseline and during week 5. We hypothesize that treatment with DTMS will be associated with significant clinical improvements in depressive and anxious symptoms, and will be well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a current major depressive disorder (according to the DSM-IV-TR) that has not improved after ≥ 1 but ≤ 5 adequate antidepressant trial(s) in the current episode
* Baseline score ≥ 15 on the QIDS-C
* Stable medication regimen (> 4 weeks)

Exclusion Criteria:

* Psychotic features in the current episode
* Lifetime history of psychotic disorders and/or bipolar I or II disorders
* Substance or alcohol abuse/dependence in the past 6 months
* Lifetime history of a major neurological disease (e.g., Parkinson's, stroke)
* Uncontrolled medical disease (e.g., cardiovascular, renal)
* Pregnancy and/or lactation
* Presence of a specific contraindication for DTMS (e.g., personal history of epilepsy, metallic head implant)
* Hearing loss
* Personal history of abnormal brain MRI findings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
21-item Hamilton Depression Rating Scale (HAM-D21) | week 5
  Response to treatment is defined as a ≥ 50% reduction in the scores of the HAM-D21. Remission is defined as a HAM-D21 score ≤ 9.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR) | week 5
  Response to treatment is defined as a ≥ 50% reduction in the scores of the QIDS-SR. Remission is defined as a QIDS-SR score ≤ 5.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo T Berlim, MD, MSc, Principal Investigator — McGill University & Douglas Mental Health University Institute
Locations (1):
- Neuromodulation Research Clinic, Douglas Mental Health University Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Isserles M, Rosenberg O, Dannon P, Levkovitz Y, Kotler M, Deutsch F, Lerer B, Zangen A. Cognitive-emotional reactivation during deep transcranial magnetic stimulation over the prefrontal cortex of depressive patients affects antidepressant outcome. J Affect Disord. 2011 Feb;128(3):235-42. doi: 10.1016/j.jad.2010.06.038. Epub 2010 Jul 21. PMID 20663568
- [Background] Levkovitz Y, Harel EV, Roth Y, Braw Y, Most D, Katz LN, Sheer A, Gersner R, Zangen A. Deep transcranial magnetic stimulation over the prefrontal cortex: evaluation of antidepressant and cognitive effects in depressive patients. Brain Stimul. 2009 Oct;2(4):188-200. doi: 10.1016/j.brs.2009.08.002. Epub 2009 Sep 16. PMID 20633419
- [Background] Levkovitz Y, Roth Y, Harel EV, Braw Y, Sheer A, Zangen A. A randomized controlled feasibility and safety study of deep transcranial magnetic stimulation. Clin Neurophysiol. 2007 Dec;118(12):2730-44. doi: 10.1016/j.clinph.2007.09.061. Epub 2007 Oct 30. PMID 17977787
- [Derived] McGirr A, Van den Eynde F, Chachamovich E, Fleck MP, Berlim MT. Personality dimensions and deep repetitive transcranial magnetic stimulation (DTMS) for treatment-resistant depression: a pilot trial on five-factor prediction of antidepressant response. Neurosci Lett. 2014 Mar 20;563:144-8. doi: 10.1016/j.neulet.2014.01.037. Epub 2014 Jan 30. PMID 24486892